CLINICAL TRIAL: NCT05561725
Title: The Impact of Perioperative Steroid Dosing on the Acute Phase Response in Adolescent Idiopathic Scoliosis
Brief Title: Perioperative Steroid Dosing on the APR in AIS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Nicholas Fletcher, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003378
Record Dates: First submitted 2022-09-20; First posted 2022-09-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Adolescent Idiopathic Scoliosis (AIS)
Keywords: Steroid; Perioperative; Posterior Spinal Fusion (PSF); Dexamethasone
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care: Control (Active Comparator): Patients will be screened for participation following indication for surgery by the treating surgeon and/or research assistant. Patients who elect to participate will then be randomized into either the dexamethasone or control groups.
  Patients in the control group will receive one 8mg dose of dexamethasone intraoperatively as per standard of care anesthesia protocols. No sham medication will be utilized for control subjects.
  Interventions: Drug: Standard of Care
- Dexamethasone (Experimental): Patients will be screened for participation following indication for surgery by the treating surgeon and/or research assistant. Patients who elect to participate will then be randomized into either the dexamethasone or control groups.
  Patients randomized to the dexamethasone cohort will be administered 8 mg of dexamethasone with 3 additional (8mg doses) administered at 8-hour intervals following surgery for a total of 4 doses.
  Interventions: Drug: Dexamethasone postoperative

INTERVENTIONS:
Drug: Dexamethasone postoperative — Patients randomized to the dexamethasone cohort will be administered 8 mg of dexamethasone with 3 additional (8mg doses) administered at 8-hour intervals following surgery for a total of 4 doses.
  All patients will undergo a standardized post-operative pathway in the hospital following surgery that has been utilized for all AIS patients at our center since 2014.
  Arms: Dexamethasone
Drug: Standard of Care — Patients in the control group will receive one 8mg dose of dexamethasone intraoperatively as per standard of care anesthesia protocols. No sham medication will be utilized for control subjects.
  All patients will undergo a standardized post-operative pathway in the hospital following surgery that has been utilized for all AIS patients at our center since 2014.
  Arms: Standard of Care: Control

SUMMARY:
The objective of this study is to perform a prospective, randomized controlled trial investigating the clinical usage of perioperative dexamethasone usage on APR activation, postoperative morphine usage, postoperative nausea, and hospital length of stay.

There will be a control control and a Dexamethasone cohort. Participants will be randomized into one of the two cohorts. Patients in the control group will receive one 8mg dose of dexamethasone intraoperatively as per standard of care anesthesia protocols. Patients randomized to the dexamethasone cohort will be administered 8 mg of dexamethasone with 3 additional doses administered at 8-hour intervals following surgery for a total of 4 doses. All study activities will tale place at Egleston during the patient's planned inpatient stay for their posterior spinal fusion.

This project has the potential to validate the utility of dexamethasone as a way to optimize postoperative care following PSF for AIS by minimizing the need for opioid medications and enhancing mobility and recovery.

DETAILED DESCRIPTION:
The objective of this study is to validate the utility of dexamethasone as a way to optimize postoperative care following PSF for AIS by minimizing the need for opioid medications and enhancing mobility and recovery.

The acute phase response (APR) is the body's response to induced tissue injury to facilitate, survive, and activate tissue repair. Posterior spinal fusion (PSF) is one source of tissue injury that has the potential to evoke an exuberant APR which can lead to a hyper-inflammatory state that can be associated with increased pain and patient morbidity. Perioperative steroid use has emerged as one potential method to minimize the activation of the APR as well as decrease postoperative pain and also narcotic utilization. However, the extent of the steroid usage on abating the activation of the APR in PSF for adolescent idiopathic scoliosis (AIS) has not been previously investigated.

The APR plays significant roles not only in the activation of inflammation postoperatively, but also for hemostasis as it helps trigger the initial fibrin clot to seal bleeding vessels.1 The inflammatory response is a later effect, that again plays a role in coagulation but also guides the transition from the survival phase response following tissue injury to the reparative phase. However, when a hyper-inflammatory state is present due to an exuberant APR activation, this transition to the reparative phase is unable to progress, resulting in a perpetuation of inflammation activation resulting in increased pain, nausea, respiratory distress, venous thromboembolism, infection, and even death.2 The ability to minimize or prevent the development of this hyper-inflammatory state holds significant implications not only for improved post-operative pain and nausea, but also for decreased postoperative complications, decreased length of stay, and resultant decreases in hospital costs.

This project has the potential to validate the utility of dexamethasone as a way to optimize postoperative care following PSF for AIS by minimizing the need for opioid medications and enhancing mobility and recovery.

ELIGIBILITY:
Inclusion Criteria:

* All patients ages 10-18 with AIS who are undergoing a PSF performed by Dr. Nicholas Fletcher at Children's Healthcare of Atlanta Egleston will be considered eligible for the study

Exclusion Criteria:

* Patients outside the inclusion parameters or with congenital or syndromic scoliosis
* Adults > 18 years old
* Pregnant women
* Prisoners
* Patients with systemic fungal infections

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Changes in C-Reactive Protein | Immediately pre-surgery, immediately post-surgery, 24 hours post-surgery, 48 hours post-surgery
  Laboratory studies to be collected will include c-reactive protein (CRP). Laboratory studies will be performed prior to surgery, post-operatively in the post-anesthesia care unit, and every morning during the in-hospital stay up to 48 hours. Studies will be analyzed in the hospital laboratory using standard sample analysis. No more than 10cc will be collected at each lab draw.
Changes in Interleukin-6 | Immediately pre-surgery, immediately post-surgery, 24 hours post-surgery, 48 hours post-surgery
  Laboratory studies to be collected will include IL-6. Laboratory studies will be performed prior to surgery, post-operatively in the post-anesthesia care unit, and every morning during the in-hospital stay up to 48 hours. Studies will be analyzed in the hospital laboratory using standard sample analysis. No more than 10cc will be collected at each lab draw.

SECONDARY OUTCOMES:
Changes in Total morphine usage | Immediately post surgery, 24 hours post-surgery and 48 hours post-surgery
  Changes in total morphine dosage (measured in morphine equivalents) during the hospital stay will be assessed and compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Fletcher, MD, Principal Investigator — Associate Professor
Locations (1):
- Children Healthcare of Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No